CLINICAL TRIAL: NCT06532409
Title: Efficacy of Oral Amoxicillin in Comparison to Intravenous Ceftriaxone in Treatment of Uncomplicated Community Acquired Pneumonia (Cap) Among Children of Age 2-5 Years of Age
Brief Title: Comparison of Efficacy of Oral Amoxicillin Versus Intravenous Ceftriaxone
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RESnTEC, Institute of Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DrAsimCHL
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Community-acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Ceftriaxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Amoxicillin (Experimental): Patients in this group will receive IV amoxicillin/CA at a dose of 100 mg per kg per day in 3 divided doses for a maximum period of 7 days.
  Interventions: Drug: Amoxicillin/CA
- IV Ceftriaxone (Experimental): Patients in this group will receive IV ceftriaxone at a dose of 75 mg per kg per day in 2 divided doses for a maximum period of 7 days.
  Interventions: Drug: IV ceftriaxone

INTERVENTIONS:
Drug: Amoxicillin/CA — Patients will receive IV amoxicillin/CA at a dose of 100 mg per kg per day in 3 divided doses for a maximum period of 7 days.
  Arms: Oral Amoxicillin
Drug: IV ceftriaxone — Patients will receive IV ceftriaxone at a dose of 75 mg per kg per day in 2 divided doses for a maximum period of 7 days.
  Arms: IV Ceftriaxone

SUMMARY:
The efficacy of oral amoxicillin is considered equal to that of ceftriaxone in community-acquired pneumonia among children. Also, there are some factors that contradict the usage of ceftriaxone, like antibiotic resistance, adverse reactions, drug cost, and the and the chances of IV trauma and infection, which is a major problem in developing countries. Therefore, this study was planned to determine the efficacy of oral amoxicillin compared with intravenous (IV) ceftriaxone in the treatment of uncomplicated ceftriaxone in community acquired pneumonia in children less than 5 years of age.

DETAILED DESCRIPTION:
The efficacy of oral amoxicillin is considered equal to that of ceftriaxone in community-acquired pneumonia among children. Also, there are some factors that contradict the usage of ceftriaxone, like antibiotic resistance, adverse reactions, drug cost, and the and the chances of IV trauma and infection, which is a major problem in developing countries. Therefore, this study was planned to determine the efficacy of oral amoxicillin compared with intravenous (IV) ceftriaxone in the treatment of uncomplicated ceftriaxone in community acquired pneumonia in children less than 5 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Children of both gender
* Aged from 2 to 5 years
* With fever >37.5 C (99.5 F)
* Will be presented with symptoms and signs of uncomplicated community acquired pneumonia

Exclusion Criteria:

* Children requiring ICU care (having cyanosis SpO2 < 85% requiring intubation within first day of admission or in state of shock)
* Children with conditions like congenital heart disease, chronic lung disease, chronic kidney disease, severe malnutrition, asthma, foreign bodies, sickle cell disease, and immunodeficiency
* Children with underlying anatomical disorders of the lung like pulmonary sequestration, tracheoesophageal fistula or congenital cystic adenoid malformation
* Children already on antibiotics
* Presence of any complication of community acquired pneumonia
* Patients having symptoms of multi-organ involvement/sepsis
* Hypersensitivity to Amoxicillin or Ceftriaxone
* Other co-existing infections like dengue, malaria, or measles

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Free from fever | 3 days
  Efficacy will be labeled yes where fever symptoms are resolved (temperature = 98.6ºF) within 3 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Children Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared with other researchers on a reasonable request.